CLINICAL TRIAL: NCT00605787
Title: TTA in Treatment of Diabetes and Dyslipidemia
Acronym: TODDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Professor Eystein S Husebye, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSD18032; NSD18032; REKIII021.01; SLV01-1232
Record Dates: First submitted 2008-01-17; First posted 2008-01-31 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: Type 2 Diabetes Mellitus; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — 1-(carboxymethylthio)tetradecane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single group (Active Comparator): Single group all treated similarly, outcome evaluated as changes within individuals during intervention
  Interventions: Drug: Tetradecylthioacetic acid (TTA)

INTERVENTIONS:
Drug: Tetradecylthioacetic acid (TTA) — 1000mg capsules once daily for 28 days

SUMMARY:
The aim of the study is to evaluate the short-term effects of tetradecylthioacetic acid (TTA) on plasma lipids and glucose in male patients with type 2 diabetes mellitus and dyslipidemia

DETAILED DESCRIPTION:
The tight linkage of obesity, insulin resistance (and frank diabetes), dyslipidemia, and hypertension has been widely observed and has been named syndrome X, or the metabolic syndrome. For many years metformin has been the only drug in clinical use with effects on insulin resistance. Recently, agonists of the peroxisome proliferator-activated receptors (PPARs) have been introduced in the treatment of type 2 diabetes. The different PPARs seem to be activated by a wide range of lipids and lipid mediators, including fatty acids. 2-tetradecylthioacetic acid (TTA) is a modified fatty acid with high affinity for the PPARgamma receptor. In animal models of obesity-related insulin resistance (obese Zucker rats and dietary manipulated Wistar rats), TTA has an insulin sensitizing effect by enhancing the insulin mediated uptake of glucose in peripheral tissues. TTA treatment promotes fatty acid catabolism in experimental animals and this could casually be linked to the improved glucose tolerance.

The protocol for the present study describes a safety assessment and therapeutic exploratory evaluation of TTA in a small subset of male type 2 diabetes patients for 4 weeks. The primary safety parameters will include general physical observational parameters, liver function test and hematological parameters. To goal is to assess the efficacy of TTA on selected metabolic parameters including fasting blood glucose and insulin, fasting plasma lipids, antioxidant status, and fibrinolytic parameters, weight, BMI and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus with HbA1c 8.0-12.0%,
* fasting S-triacylglycerol 2.0-10.0 mmol/L,
* body mass index 25-40 kg/m2 and/or waist/hip ratio > 0.90.

Exclusion Criteria:

* fasting total cholesterol >10 mmol/L,
* blood pressure 170/110 mmHg
* other significant disease
* Use of any corticosteroid, anticoagulant or lipid-lowering drug 2 weeks prior to inclusion.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2002-01; Primary Completion 2003-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plasma lipids | -28 days, baseline, 14 and 28 days of TTA

SECONDARY OUTCOMES:
Plasma glucose | -28 days, baseline, 14 and 28 days of TTA
Safety blood parameters | -28 days, baseline, 14 and 28 days of TTA

CONTACTS AND LOCATIONS:
Overall Officials: Eystein S Husebye, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Bergen, Norway

REFERENCES:
- [Derived] Lovas K, Rost TH, Skorve J, Ulvik RJ, Gudbrandsen OA, Bohov P, Wensaas AJ, Rustan AC, Berge RK, Husebye ES. Tetradecylthioacetic acid attenuates dyslipidaemia in male patients with type 2 diabetes mellitus, possibly by dual PPAR-alpha/delta activation and increased mitochondrial fatty acid oxidation. Diabetes Obes Metab. 2009 Apr;11(4):304-14. doi: 10.1111/j.1463-1326.2008.00958.x. PMID 19267708